CLINICAL TRIAL: NCT01230073
Title: Treatment Satisfaction With Remote Monitoring in Implantable Cardioverter Defibrillator Recipients
Brief Title: Treatment Satisfaction in Implantable Cardioverter Defibrillator Recipients
Acronym: SAN REMO 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-004
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Improvement of Treatment Satisfaction
Keywords: ICD; Home-Monitoring; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICD traditional follow-up (Active Comparator): ICD with traditional follow-up in the outpatient clinic
  Interventions: Device: Home-Monitoring; Device: Follow-up by Home-Monitoring
- Home-Monitoring (Active Comparator): Home-Monitoring
  Interventions: Device: Home-Monitoring; Device: Follow-up by Home-Monitoring

INTERVENTIONS:
Device: Home-Monitoring — Home-Monitoring
Device: Follow-up by Home-Monitoring — Follow-up by Home-Monitoring

SUMMARY:
Remote monitoring of implantable cardioverter defibrillators (ICD) is a promising new development in ICD therapy and has been shown to be technically feasible and safe.While data on safety and feasibility of remote monitoring are in favour of this technology, patients´ treatment satisfaction has not been sufficiently investigated. To date, there is only one small, non-randomised study investigating patients´ treatment satisfaction in highly selected and highly motivated patients at the time of implantation and 12 months thereafter7. Therefore, the aim of the San Remo Trial is to investigate factors that are associated with patients´ willingness to accept the new method of follow-up on a broad basis of ICD recipients and to determine their treatment satisfaction with ICD therapy in a randomised, prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication according to current national or international guidelines
* Patient available for follow-up during study period

Exclusion Criteria:

* Clinically unstable medical conditions that require regular outpatient clinic follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2014-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction with ICD therapy and follow-up | 12 months

SECONDARY OUTCOMES:
Number of healthcare consultations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kolb Christof, Principal Investigator — Deutsches Herzzentrum
Locations (1):
- Deutsches Hezzentrum, München, Bavaria, Germany